CLINICAL TRIAL: NCT05839353
Title: Evaluation of the Effect of Training in the SBAR (Situation Background Assessment Recommendation) Tool on the Feeling of Self-efficacy of Carers of Patients With Lung Cancer in the Face of a Situation of Simulated Respiratory Distress.
Brief Title: Evaluation of the Effect of Training in the Situation Background Assessment Recommendation (SBAR) Tool on the Feeling of Self-efficacy of Carers of Patients With Lung Cancer in the Face of a Situation of Simulated Respiratory Distress.
Acronym: SAECURE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/CHU/20; 2023-A00914-41 (Other: id-RCB)
Record Dates: First submitted 2023-04-20; First posted 2023-05-03 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Caregivers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- simulated training by Serious Game (SG): Simulated training (by SG) for the use of the SBAR tool associated with the usual instructions issued in routine care, on the management of dyspnea
  Interventions: Other: SBAR training by serious game
- usual instructions issued in routine care: Usual instructions issued in routine care, on the management of dyspnea

INTERVENTIONS:
Other: SBAR training by serious game — SBAR training by serious game
  Groups: simulated training by Serious Game (SG)

SUMMARY:
Dyspnea is defined as a subjective feeling of discomfort in breathing. In respiratory pathologies, dyspnea can be indicative of lung cancer or its aggravation, or even be the most important symptom of the end of life. The prevalence of dyspnea is high in patients with lung cancer, ranging from 50 to 87%. Dyspnea can exacerbate at any time in the course of care for the patient with lung cancer, causing respiratory distress or Acute Respiratory Failure (ARF) and putting the prognosis at stake. ARF justifies urgent and effective care, and in pre-hospital, it is based on the call to the Emergency Medical Aid Service (SAMU). The communication of information on the patient's condition in ARF to the SAMU must be as clear and precise as possible in order to avoid medical errors, inappropriate decisions and therefore a loss of opportunity for the patient. In Oncology, caregivers often assume the role of "decision maker" and provide monitoring and assessment of symptoms, including dyspnea.

A qualitative study on the experience of caregivers during dyspnea occurring in patients with lung cancer or obstructive bronchopneumopathy revealed an altered emotional state of caregivers, such as anxiety, stress and feeling of helplessness, especially when respiratory deterioration occurs suddenly at night. The unmet need for information could compromise the sense of self-efficacy among caregivers.

In this context of monitoring symptoms in lung cancer at home, caregivers are the first witnesses of respiratory distress in their loved ones. However, faced with the sudden deterioration of breathing, they risk forgetting to communicate essential information when calling the SAMU. Since 2014, the High Authority for Health (HAS) has been recommending the use of the SBAR tool (Situation, Background, Assessment Recommendation) to facilitate communication between professionals. Its effectiveness has been proven both in improving knowledge and in the quality of communication. This is why training in the use of the SBAR (Situation, Background, Assessment Recommendation) tool could be extrapolated to caregivers with regard to the responsibilities they must assume in the management of home care, including lung cancer to deal with respiratory distress.The Serious Game (SG) is an innovative educational tool adapted to training in the field of health.It is an interactive web-based software allowing the repetitive training of medical procedures in a virtual environment, in the form of video games for active, experiential and problem-based learning, without the need to involve patients and therefore without risk.The aim of the research is to provide training in the SBAR (Situation, Background, Assessment Recommendation) tool in the form of a Serious Game for carers of patients with lung cancer in order to improve the feeling of self-efficacy in the management of respiratory distress at home.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Designated as a resource person by a patient newly diagnosed with lung cancer and receiving their first course of anti-cancer treatment (chemotherapy, hormone therapy or targeted therapy)
* Providing daily unpaid technical, psychological and social assistance
* Having given free, informed, express oral consent

Exclusion Criteria:

* Person deprived of liberty by judicial or administrative decision, and person subject to legal protection (guardianship or curators)
* Having a cancerous pathology
* Illiterate
* Do not have access to computer equipment (computer, tablet or smart phone)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Designated as a resource person by a patient newly diagnosed with lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Effect of training in the SBAR tool by serious game on the feeling of self-efficacy of carers of patients with lung cancer in the face of a situation of simulated respiratory distress. | 28 days
  Generalized Self-Efficacy (GSE) scale _ 10 question / minimum value = 10 ; maximum value = 40 / Higher scores mean a better outcome (high sense of self-efficacy)

SECONDARY OUTCOMES:
Effect of training in the SBAR tool by serious game on anxiety | 28 and 90 days
  Hospital Anxiety and Depression Scale (HADS) _ 14 question / minimum value = 7 or mean ; maximum value > 11 / Higher scores mean a worse outcome (high anxiety and depression)
Effect of training in the SBAR tool by serious game on stress | 28 and 90 days
  Perceived Stress Scale-10 (PSS 10) _ 10 question / minimum value = 0 ; maximum value = 40 / Higher scores mean a worse outcome (high stress)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle REYNAUD, Principal Investigator — CHU Reunion Island
Locations (1):
- Reunion Island University Hospital, Saint-Pierre, France

IPD SHARING:
Plan to Share IPD: No